CLINICAL TRIAL: NCT07320521
Title: A Phase I Study to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]HRS-8080 in Healthy Chinese Postmenopausal Female Subjects.
Brief Title: A Study to Assess the Mass Balance of [14C]HRS-8080 in Healthy Chinese Postmenopausal Female Subjects.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8080-103
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]HRS-8080 Group (Experimental)
  Interventions: Drug: [14C]HRS-8080

INTERVENTIONS:
Drug: [14C]HRS-8080 — Subjects will receive single dose of orally [14C]HRS-8080.

SUMMARY:
This single-part, healthy volunteer study will try to identify how the test medicine is taken up, broken down and removed from the body. To help investigate this, the test medicine is radiolabelled, which means that the test medicine has a radioactive component (carbon-14) which helps us to track where the test medicine is in the body. The safety and tolerability of the test medicine will also be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy postmenopausal female.
2. Body weight must be ≥45 kg at screening, and Body Mass Index (BMI) must be within the range of 19 kg/m² to 26 kg/m² (inclusive).
3. The subject must have regular bowel movements.

Exclusion Criteria:

1. Any clinically significant disease or disorder that the researcher believes may pose a risk to the researcher due to participation in the study, or may affect the research results.
2. Have participated in blood donation within 3 months prior to screening, with a blood donation volume of ≥400 mL or a blood loss of ≥400 mL; Have participated in blood donation within one month and donated at least 200 mL of blood or lost at least 200 mL of blood; Those who receive blood transfusion within one month or plan to donate blood within three months after the end of this trial.
3. Having taken any clinical trial drug or participated in any drug clinical trial within the three months prior to the screening period.
4. Those who have received a vaccine within one month before screening or plan to receive a vaccine during the trial period.
5. People with allergic constitutions, such as those with a known history of allergy to two or more substances; Or those who, as determined by the researchers, may be allergic to the investigational drug or its excipients.
6. Those with a history of fainting at the sight of needles or blood may have difficulty in blood collection or cannot tolerate venipuncture for blood collection.
7. Workers engaged in work that requires long-term exposure to radioactive conditions; Or those who have had significant radioactive exposure within one year prior to the test or have participated in radioactive drug labeling tests.
8. Those who show abnormal results through comprehensive physical examination, vital signs, laboratory tests, 12-lead electrocardiogram, chest X-ray, digital rectal examination, and abdominal B-ultrasound, and are determined by the researcher to have clinical significance.
9. Sex hormones: Those with abnormal tests for luteinizing hormone (LH), progesterone (P), testosterone (T), and prolactin (PRL), and who are determined by the researcher to have clinical significance.
10. Excessive drinking or frequent alcohol consumption within the six months prior to the screening period, that is, consuming more than 14 units of alcohol per week (1 unit =360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine); Or the result of the alcohol breath test during the screening period is ≥20 mg/dl; Or those who are unable to quit alcohol during the trial period.
11. Those who smoked more than five cigarettes per day or habitually used nicotine-containing products in the three months prior to the screening period; Or those who are unable to withdraw during the trial period.
12. Abuse of drugs or use of soft drugs (such as marijuana) in the three months prior to the screening period or use of hard drugs (such as cocaine, amphetamines, etc.) in the year prior to the screening period; Or positive urine drug abuse (drug) test during the screening period.
13. Those who habitually consume grapefruit juice or excessive amounts of tea, coffee and/or caffeinated beverages and are unable to quit during the trial period.
14. Any significant abnormalities in the 12-lead electrocardiogram during screening were considered clinically significant by the researchers.
15. Those with any history of serious clinical diseases or diseases or conditions that the researcher believes may affect the trial results, such as a history of gastrointestinal, liver or kidney diseases or current existence of such diseases, or any diseases known to interfere with drug absorption, distribution, metabolism or excretion.
16. Those who test positive for any one of hepatitis B surface antigen or hepatitis B e antigen, hepatitis C virus antibody, Treponema pallidum antibody, or the combined test of human immunodeficiency virus antigen/antibody.
17. There was evidence of renal insufficiency during screening.
18. Those who have undergone major surgery within 6 months prior to the screening period or whose surgical incisions have not fully healed; Major surgeries include but are not limited to those with significant bleeding risks, prolonged general anesthesia periods, or incision biopsies or obvious traumatic injuries.
19. Hemorrhoids or perianal diseases accompanied by regular or ongoing bleeding during defecation; Subjects who are unable to swallow, or have a history of gastrointestinal dysfunction such as irritable bowel syndrome, inflammatory bowel disease, or have undergone surgeries like gastrectomy, which the researchers determine may affect drug absorption, as well as those with habitual constipation or diarrhea.
20. Any drugs that inhibit or induce the activity of liver drug-metabolizing enzymes or transporters have been used within 30 days prior to screening.
21. In the 14 days prior to screening or currently using any prescription drugs, over-the-counter drugs, vitamin products, health supplements or Chinese herbal medicines, etc., unless it has been evaluated that the use of such drugs will not interfere with the research objectives and will not endanger the safety of the subjects.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The cumulative amount of HRS-8080 excreted. | 0 hour to 360 hours.
Percentage of parent drug and its metabolite(s) relative to total radioactive exposure in plasma. | 0 hour to 360 hours.
Percentage of administered dose excreted as parent drug and its metabolite(s) in urine. | 0 hour to 360 hours.
Percentage of administered dose excreted as parent drug and its metabolite(s) in feces. | 0 hour to 360 hours.
Maximum concentration (Cmax). | 0 hour to 336 hours.
  Pharmacokinetic parameters for total radioactivity in plasma.
Time of maximum concentration (Tmax). | 0 hour to 336 hours.
  Pharmacokinetic parameters for total radioactivity in plasma.
Area under the concentration-time curve (AUC). | 0 hour to 336 hours.
  Pharmacokinetic parameters for total radioactivity in plasma.
Elimination half-life (t1/2). | 0 hour to 336 hours.
  Pharmacokinetic parameters for total radioactivity in plasma.
Apparent clearance (CL/F). | 0 hour to 336 hours.
  Pharmacokinetic parameters for total radioactivity in plasma.
Apparent volume of distribution (Vz/F). | 0 hour to 336 hours.
  Pharmacokinetic parameters for total radioactivity in plasma.
Ratio of total radioactivity in whole blood to plasma. | 0 hour to 360 hours.

SECONDARY OUTCOMES:
Maximum concentration (Cmax). | 0 hour to 336 hours.
  Pharmacokinetic parameters for HRS-8080 and its metabolite(s) in plasma.
Time of maximum concentration (Tmax). | 0 hour to 336 hours.
  Pharmacokinetic parameters for HRS-8080 and its metabolite(s) in plasma.
Area under the concentration-time curve (AUC). | 0 hour to 336 hours.
  Pharmacokinetic parameters for HRS-8080 and its metabolite(s) in plasma.
Elimination half-life (t1/2). | 0 hour to 336 hours.
  Pharmacokinetic parameters for HRS-8080 and its metabolite(s) in plasma.
Apparent clearance (CL/F). | 0 hour to 336 hours.
  Pharmacokinetic parameters for HRS-8080 and its metabolite(s) in plasma.
Apparent volume of distribution (Vz/F). | 0 hour to 336 hours.
  Pharmacokinetic parameters for HRS-8080 and its metabolite(s) in plasma.
Adverse events (AEs). | Day -7 to Day 23.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided